CLINICAL TRIAL: NCT06758466
Title: A Prospective Randomized Controlled Trial Comparing Bipolar TURP and Bipolar Enucleation of the Prostate for Benign Prostatic Hyperplasia (BPH) With Prostate Volumes Between 30-80 Grams
Brief Title: Bipolar TURP Versus Bipolar Enucleation for BPH Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Samer Morsy, Associate Professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kasr Alainy- Cairo University
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH - Bipolar- TURP - Enucleation
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar enucleation (Active Comparator)
  Interventions: Procedure: Prostate surgery
- Bipolar resection (Active Comparator)
  Interventions: Procedure: Prostate surgery

INTERVENTIONS:
Procedure: Prostate surgery — Prostate removal

SUMMARY:
To compare the surgical outcomes at 12 months post-surgery between Bipolar TURP and BipoLEP in men with BPH and prostate volumes between 30-80 grams.

DETAILED DESCRIPTION:
Create a research protocol in a prospective study to compare bipolar transurethral resection of prostate vs bipolar enucleation of prostate between 30 and 80 gm in management of BPH

Okay, here's a detailed research protocol for a prospective study comparing Bipolar Transurethral Resection of the Prostate (TURP) and Bipolar Enucleation of the Prostate (BipoLEP) for BPH, specifically focusing on prostates between 30-80 grams:

Study Title: A Prospective Randomized Controlled Trial Comparing Bipolar TURP and Bipolar Enucleation of the Prostate for Benign Prostatic Hyperplasia (BPH) with Prostate Volumes between 30-80 grams

1. Introduction

Background: Briefly introduce Benign Prostatic Hyperplasia (BPH), its prevalence, and the associated lower urinary tract symptoms (LUTS). Highlight the common surgical interventions: TURP and, more recently, enucleation techniques.

Problem Statement: State that while both bipolar TURP and BipoLEP are established treatments, there's a need for a direct comparison, especially for moderate-sized prostates (30-80g). There's an ongoing debate regarding which approach offers superior outcomes and a better balance of efficacy and safety.

Rationale: Explain why this study is necessary. This can be because there is limited direct

Primary Objective: To compare the International Prostate Symptom Score (IPSS) at 12 months post-surgery between Bipolar TURP and BipoLEP in men with BPH and prostate volumes between 30-80 grams.

Secondary Objectives:

To compare perioperative outcomes including:

Operative time (minutes)

Catheterization time (days)

Length of hospital stay (days)

Blood loss (change in hemoglobin)

Requirement of blood transfusion

Incidence of perioperative complications (e.g., TUR syndrome, bleeding, infection, clot retention)

To compare postoperative functional outcomes including:

Peak urinary flow rate (Qmax) at 3, 6, and 12 months

Post-void residual (PVR) volume at 3, 6, and 12 months

Quality of life (QoL) using a validated questionnaire at 3, 6, and 12 months

To compare the incidence of postoperative complications including:

Urinary tract infection (UTI)

Urinary incontinence (UI)

Urethral stricture

Bladder neck contracture

Need for re-operation within 12 months.

To compare overall patient satisfaction using a visual analog scale (VAS) at 3, 6, and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 45-80 years diagnosed with symptomatic BPH.
* Prostate volume between 30-80 grams as determined by transrectal ultrasound (TRUS) performed within 4 weeks before randomization.
* Moderate to severe LUTS with an IPSS of ≥ 8.
* Failure of medical management.
* Patients able to provide written informed consent.

Exclusion Criteria:

* History of prostate cancer.
* History of previous prostate surgery (including any procedure for BPH or prostate cancer).
* History of urethral stricture or bladder neck contracture.
* Neurogenic bladder dysfunction.
* Significant coagulopathy.
* Uncontrolled urinary tract infection.
* Patient on anticoagulant medication.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — BPH
Enrollment: 180 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 12 months
Qmax | 12 months

SECONDARY OUTCOMES:
PVR | 12 months
Complications | 12 months